CLINICAL TRIAL: NCT00433472
Title: Effect of RSR13 on T2 and T2* Cranial MRI Images: An Imaging Companion Study to NABTT 9806
Brief Title: MRI in Evaluating the Effect of Efaproxiral on the Brain in Patients With Recurrent or Progressive Glioma Enrolled on Clinical Trial NABTT-9806
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough interest
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Joy Fisher, ABTC Consortium
Purpose: Diagnostic
Other Study IDs: NABTT-2002 CDR0000274785; U01CA062475 (NIH); P30CA006973 (NIH); NABTT-2002; JHOC-NABTT-2002; ALLOS-RSR13CT-001i
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult anaplastic astrocytoma; recurrent adult brain tumor; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Glioblastoma; Astrocytoma; Brain Neoplasms; Gliosarcoma | interventions — Magnetic Resonance Imaging

ARMS (1):
- MRI - (Other): MRI scan to be complete to look at RSR13 on measurement of T2 and T2* on MRI
  Procedure/surgery magnetic resonance imaging (MRI)
  Interventions: Device: magnetic resonance imaging (MRI)

INTERVENTIONS:
Device: magnetic resonance imaging (MRI) — MRI scan to be complete to look at RSR13 on measurement of T2 and T2* on MRI
  Other Names: MRI

SUMMARY:
RATIONALE: Diagnostic procedures, such as MRI, may help doctors learn how efaproxiral works in the brain and help plan the best treatment.

PURPOSE: This clinical trial is using MRI to evaluate the effect of efaproxiral on the brain in patients with recurrent or progressive glioma receiving treatment on clinical trial NABTT-9806.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether efaproxiral has a measurable effect on the brain as shown by T2 and/or T2* MRI in patients with recurrent or progressive malignant glioma enrolled on NABTT-9806.
* Determine predicted oxygenation changes based on observed T2 MRI changes in these patients.
* Determine the effects of this drug on T2 and T2* MRI relaxation times of normal areas of the brain in these patients.
* Determine baseline oxygen extraction ratios in tumors of patients treated with this drug.
* Determine whether administration of this drug reveals any new tumor- or non-tumor-related abnormalities on T2 and T2* MRI in these patients.

OUTLINE: This is an open-label, multicenter, pilot study.

Patients receive efaproxiral and carmustine on clinical trial NABTT-9806. During any one course of treatment on that study, patients undergo MRI before oxygen administration (baseline), before efaproxiral infusion, and then every 5 minutes until 1 hour after efaproxiral and carmustine treatment. Data is evaluated for extent and intensity of T2/T2* changes and oxygen concentration changes in both abnormal and normal brain.

PROJECTED ACCRUAL: A total of 15-48 patients will be accrued for this study within 12-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Recurrent or progressive glioma
* Currently enrolled on clinical trial NABTT-9806

PATIENT CHARACTERISTICS:

* No severe claustrophobia
* No cardiac pacemaker
* No MRI-incompatible metallic implant

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Measurable effect of efaproxiral on the brain as measured by T2 and/or T2* MRI
Predicted oxygenation changes based on observed T2 MRI changes
Effects of efaproxiral on T2 and T2* MRI relaxation times of normal areas of the brain
Baseline oxygen extraction ratios in tumors
New tumor- or non-tumor-related abnormalities on T2 and T2* MRI

CONTACTS AND LOCATIONS:
Overall Officials: Larry Kleinberg, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins